CLINICAL TRIAL: NCT06391034
Title: A Phase 2 Study of Magnetic Resonance (MR) Imaging With Hyperpolarized 13C-Pyruvate +/- 13C,15N-Urea in Patients With Prostate Cancer Undergoing Radiation Therapy
Brief Title: Magnetic Resonance (MR) Imaging With Hyperpolarized 13C-Pyruvate +/- 13C,15N-Urea in Patients With Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Bok, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Bok, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24922; 5R01CA238379 (NIH); NCI-2024-03775 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Imaging Studies; Hyperpolarized 13C-Pyruvate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Image Optimization Group (Experimental): Participants will undergo Hyperpolarized 13C-Pyruvate +/- 13C,15N-Urea imaging as part of a multi-parametric magnetic resonance imaging (mpMRI) exam, with the primary objective of optimizing imaging sequences and techniques to maximize signal-to-noise ratio of imaging modality.
  Interventions: Drug: hyperpolarized pyruvate +/-urea (13C/15N); Procedure: Multi-parametric magnetic resonance imaging (mpMRI)
- Part 2A: Prospective imaging (External beam radiotherapy (EBRT) Participants) (Experimental): Participants with pre-planned, non-interventional stereotactic body radiotherapy (EBRT) will undergo an HP Pyruvate +/-Urea mpMRI exam at baseline, at 3 months post-EBRT treatment and at 1yr post-treatment.
  Interventions: Drug: hyperpolarized pyruvate +/-urea (13C/15N); Radiation: Non-investigational External beam radiotherapy (EBRT); Procedure: Multi-parametric magnetic resonance imaging (mpMRI)
- Part 2B: Prospective imaging (High-risk localized prostate cancer) (Experimental): Participants with with high-risk localized prostate cancer and have pre-planned, non-interventional primary radiation therapy (RT) with concurrent, systemic, non-interventional hormone therapy will undergo HP Pyruvate+/-Urea mpMRI at baseline prior to the start of systemic hormone therapy, 4-12 weeks after the initiation of systemic hormone therapy (prior to radiation therapy), at 3 months post-radiation therapy, and at +1yr post-radiation therapy.
  Interventions: Drug: hyperpolarized pyruvate +/-urea (13C/15N); Procedure: Radiotherapy (RT); Procedure: Multi-parametric magnetic resonance imaging (mpMRI); Biological: Non-interventional hormone therapy
- Part 3: EBRT participants at time of biochemical recurrence (BCR) (Experimental): Evaluable EBRT participants who undergo HP Pyruvate +/-Urea mpMRI at time of biochemical failure, followed by magnetic resonance (MR) / ultrasound (US) fusion-guided prostate biopsy within 12 weeks following baseline MR exam. Participants in this group have the option of undergoing a follow up HP Pyruvate +/-Urea MR exam 6-15 months following the baseline scan, to evaluate for any interval change.
  Interventions: Drug: hyperpolarized pyruvate +/-urea (13C/15N); Radiation: Non-investigational External beam radiotherapy (EBRT); Procedure: Multi-parametric magnetic resonance imaging (mpMRI); Procedure: Prostate Biopsy

INTERVENTIONS:
Drug: hyperpolarized pyruvate +/-urea (13C/15N) — Given IV
  Other Names: 13C-Pyruvate,15N-urea
Radiation: Non-investigational External beam radiotherapy (EBRT) — External beam radiotherapy given outside of this study
  Other Names: EBRT
  Arms: Part 2A: Prospective imaging (External beam radiotherapy (EBRT) Participants); Part 3: EBRT participants at time of biochemical recurrence (BCR)
Procedure: Radiotherapy (RT) — Radiation therapy given outside of this study
  Other Names: RT
  Arms: Part 2B: Prospective imaging (High-risk localized prostate cancer)
Procedure: Multi-parametric magnetic resonance imaging (mpMRI) — Imaging scan
  Other Names: mpMRI
Biological: Non-interventional hormone therapy — Therapy given outside of this study as part of standard of care
  Other Names: Non-interventional, systemic hormone therapy
  Arms: Part 2B: Prospective imaging (High-risk localized prostate cancer)
Procedure: Prostate Biopsy — Biopsies may be taken from Trans-rectal ultrasound (TRUS) -visible lesion at the urologist's discretion
  Other Names: Biopsy
  Arms: Part 3: EBRT participants at time of biochemical recurrence (BCR)

SUMMARY:
This is a Phase 2 clinical study of hyperpolarized (HP) 13C-pyruvate (13C), 15N-urea (13C,15N) metabolic MR imaging in prostate cancer patients who are undergoing or have received radiation therapy for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Part 1: To Optimize the imaging sequences that maximize signal-to-noise ratio (SNR) and intra-tumoral kPL and kPG in regions of tumor vs. adjacent benign tissue as assessed by mpMRI imaging characteristics.

II. Part 2A To perform HP 13C-MRI and measure the changes in tumoral kPL and kPG.

III. Part 2B: To perform HP 13C-MRI and study the metabolic effects (changes in tumor kPL and kPG).

IV. Part 3: To perform HP 13C-MRI at time of Biochemical Failure and measure tumoral kPL and kPG, in previously external beam radiation therapy (EBRT) treated patients.

SECONDARY OBJECTIVES:

I. To evaluate the intra-patient variability in intra-tumoral kPL and kPG with repeated dose studies (Part 1, 2 & 3).

II. To determine the association between peak intra-tumoral kPL observed on baseline imaging with serum PSA. (Part 2 & 3).

III. To determine the association between changes in intra-tumor kPL after 4-12 weeks of systemic hormone therapy and PSA response (Part 2B).

IV. To compare and contrast intra-tumoral kPL and kPG with Prostate Imaging Reporting and Data System (PI-RADS) version 2 and individual mpMRI parameters including apparent diffusion coefficient (ADC) on diffusion-weighted imaging (Part 1, 2 & 3).

V. To describe the frequency of up-grading of tumor with MR/US-guided fusion biopsy obtained following baseline HP-MRI exam. (Part 3).

VI. To further characterize the safety profile of HP C-13 pyruvate injections (Part 1, 2 & 3).

VII. For patients imaged with HP 13C-MRI at time of biochemical failure post-EBRT, correlate peak intra-tumoral kPL and kPG with radiotherapy dose distributions from EBRT course (Part 3).

VIII. For studies incorporating HP 13C-urea, the baseline and the on-treatment changes in urea AUC parameter will be measured and compared to kPL endpoints of the same lesions (Part 1, 2 & 3).

OUTLINE:

The study is divided into 3 parts. Part 1: Participants undergo imaging as part of a multi-parametric magnetic resonance imaging (mpMRI) exam to determine exact parameters for imaging.

Part 2A: Participants planned for external beam radiotherapy (EBRT) Part 2B: Participants with high-risk localized prostate cancer planned to receive primary radiation therapy with concurrent systemic hormone therapy Part 3: Evaluable EBRT participants scanned at time of biochemical failure and MR/US fusion-guided prostate biopsy within 12 weeks. Participants have the option of undergoing a follow up HP Pyruvate +/- Urea MR exam 6-15 months following the baseline scan.

All participants will receive a scan at baseline and other procedures may be performed as part of routine, non-interventional standard of care at the time of biochemical failure, including serial prostate-specific antigen (PSA) monitoring and gene expression profiling of tumor tissue. Participants will be followed for 24 months after last procedure or removal from study, or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have biopsy-proven adenocarcinoma of the prostate, as determined by medical chart review.
2. For:

   1. Part 1: Participants post-radiation therapy or currently considering EBRT.
   2. Part 2A: Participants currently scheduled for or considering EBRT (no neo-adjuvant therapy planned).
   3. Part 2B: Participants currently scheduled for or considering EBRT and neo-adjuvant therapy is planned. The participant has biopsy-proven adenocarcinoma of the prostate with high-risk disease, defined by the presence of at least two of following criteria: a tumor stage of T3 or T4, a Gleason score of 8 to 10, or a PSA level ≥40 ng/mL) and the participant must be planning to receive androgen deprivation therapy (ADT) with an Luteinizing hormone-releasing hormone (LHRH) agonist or antagonist. The addition of an androgen-receptor (AR) signaling inhibitor (e.g., abiraterone, bicalutamide,apalutamide, enzalutamide or darolutamide) will be allowed.
   4. Part 3: Participants who have previously received radiation treatment to the prostate and are exhibiting signs of biochemical failure, with planned fusion biopsy within 12 weeks following completion of baseline HP 13C pyruvate +/-urea mpMRI.
3. Participant is able and willing to comply with study procedures and provide signed and dated informed consent.
4. Eastern Cooperative Oncology Group (ECOG) performance status <= 1.
5. Age >= 18 years old at time of study entry.
6. Ability to understand and the willingness to sign a written informed consent document.
7. Demonstrates adequate organ function as defined below:

   1. White Blood Cell count (WBC) >=4000 cells/μL.
   2. Hemoglobin ≥9.0 gm/dL.
   3. Platelets ≥75,000 cells/μL.
   4. Renal Function > 30 Epithelial Growth Factor Receptor (eGFR).

Exclusion Criteria:

1. Evidence of pelvic regional or distant metastatic disease on conventional imaging (MRI, computed tomography or whole body bone scan) or prostate-specific membrane antigen (PSMA) Positron Emission Tomography (PET) imaging. PSMA-avid lymph nodes confined to the pelvis will be allowed if <1 centimeter (cm).
2. Prostate biopsy performed within 14 days prior to baseline C-13 HP pyruvate MRI.
3. Poorly controlled hypertension, with blood pressure at study entry > 160 mm Hg systolic or > 100 mm Hg diastolic. Treatment with anti-hypertensives and re-screening is permitted.
4. Contraindication to or inability to tolerate MRI with endorectal coil (e.g. severe claustrophobia, presence of cardiac pacemaker, aneurysm clip, severe or painful hemorrhoids, rectal stricture).
5. Congestive heart failure with New York Heart Association (NYHA) status >= 2.
6. History of clinically significant ECG abnormality, including QT prolongation, a family history of prolonged QT interval syndrome or myocardial infarction within 6 months of study entry.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Signal-to-noise ratio (Part 1) | Day of MR imaging (1 day)
  A signal-to-noise ratio is defined as a MR/spectroscopy parameter, consisting of the HP C13-Pyruvate or Lactate signal (peak) relative to background noise level (baseline) in MRI spectra of the tissue.
Mean HP 13C-pyruvate to lactate metabolic rate of conversion (kPL) over time (Part 2A) | Up to 24 months
  The mean percent change in tumoral kPL between baseline and 1-year post-EBRT will be reported.
Mean HP 13C-pyruvate to glutamate metabolic rate of conversion (kPG) over time (Part 2A) | Up to 24 months
  The mean percent change in tumoral kPG between baseline and 1-year post-EBRT will be reported.
Mean change in on-treatment kPL over time (Part 2B) | Up to 24 months
  Mean percent change in tumoral kPL for participants receiving systemic hormone therapy between baseline and 1 -year post-EBRT will be reported.
Mean change in on-treatment kPG over time (Part 2B) | Up to 24 months
  Mean percent change in tumoral kPG for participants receiving systemic hormone therapy between baseline and 1 -year post-EBRT will be reported.
Mean kPL at time of biochemical failure (Part 3) | Up to 24 months
  The mean kPL for participants with biochemical failure will be reported.
Mean kPG at time of biochemical failure (Part 3) | Up to 24 months
  The mean kPG for participants with biochemical failure will be reported.

SECONDARY OUTCOMES:
Intra-patient variability of kPL | Up to 12 months
  Intra-patient variability in the kPL will be summarized by the intraclass correlation and presented with a 90% confidence interval when multiple HP-MRI scans are obtained for a participant.
Intra-patient variability of kPG | Up to 12 months
  Intra-patient variability in the kPG will be summarized by the intraclass correlation and presented with a 90% confidence interval when multiple HP-MRI scans are obtained for a participant.
Mean intra-tumoral kPL above and below the median PSA (Parts 2-3) and the mean serum PSA | Up to 24 months
  The study cohort will be dichotomized by mean intra-tumoral kPL obtained at baseline with median serum PSA and will be compared between the two dichotomized subgroups using Mann-Whitney test.
Correlation of kPL with Prostate Imaging Reporting and Data System (PI-RADS) version 2 classification score | Up to 24 months
  Spearman's rank order correlation coefficient will be used to determine the relationship between kPL with PI-RADS version 2 classification score (1 through 5; PI-RADS 1 - Very low (clinically significant cancer is highly unlikely to be present) PI-RADS 2 - Low (clinically significant cancer is unlikely to be present)). The Spearman's correlation coefficient (rs) measures the strength and direction of association between two variables. The Spearman correlation coefficient, rs, can take values from +1 to -1 where a value of +1 indicates a perfect association, an rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association.
Correlation of kPG with PI-RADS version 2 classification score | Up to 24 months
  Spearman's rank order correlation coefficient will be used to determine the relationship between kPL with PI-RADS version 2 classification score (1 through 5; PI-RADS 1 - Very low (clinically significant cancer is highly unlikely to be present) PI-RADS 2 - Low (clinically significant cancer is unlikely to be present)). The Spearman's correlation coefficient (rs) measures the strength and direction of association between two variables. The Spearman correlation coefficient, rs, can take values from +1 to -1 where a value of +1 indicates a perfect association, an rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association.
Proportion of participants with concordant mismatch of low HP 13C-urea perfusion (ureaAUC) | Up to 24 months
  A secondary endpoint will be to identify concordant mismatch of low HP 13C-urea perfusion (ureaAUC) in lesions assessed for kPL.
Mean percent change in kPL over time for participants with optional scan | Up to 24 months
  For the subset of participants who undergo optional follow up MR scan following baseline MRI, the mean percent change from baseline in kPL will be descriptively reported using summary statistics.
Number of participants with reported treatment-related adverse events | From start of HP 13C-pyruvate MR imaging to 20 minutes after the procedure for all scans
  The incidence of adverse events as graded by Common Toxicity Criteria version 5.0 will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bok, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No